CLINICAL TRIAL: NCT06754059
Title: A Single-arm, Multicenter, Real-world Observational Study of Pyrotinib Combined With Trastuzumab for Maintenance Therapy After First-line TH (P) Therapy for HER2+ABC
Brief Title: Pyrotinib Combined With Trastuzumab for Maintenance Therapy After First-line TH (P) Therapy for HER2+ABC
Status: Recruiting | Type: Observational
Sponsor: zhangjie (Other)
Responsible Party: Sponsor-Investigator, zhangjie, Clinical Professor, Fujian Medical University Union Hospital
Organization: Fujian Medical University Union Hospital (Other)
Other Study IDs: Fujian union BC-001
Record Dates: First submitted 2024-12-23; First posted 2024-12-31 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: HER2-positive Breast Cancer
MeSH Terms: interventions — pyrotinib

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pyrotinib: In this study, after at least 4 cycles of taxoid chemotherapy combined with trastuzumab ± pertuzumab, the evaluation result reached SD, CR or PR, and capecitabine combined with pyrotinib + trastuzumab was given successively in the later period(capecitabine was used for 4-6 cycles
  Interventions: Drug: Pyrotinib

INTERVENTIONS:
Drug: Pyrotinib — In this study, after at least 4 cycles of taxoid chemotherapy combined with trastuzumab ± pertuzumab, the evaluation result reached SD, CR or PR, and capecitabine combined with pyrotinib + trastuzumab was given successively in the later period (capecitabine was used for 4-6 cycles

SUMMARY:
A single-arm, multicenter, real-world observational study of pyrotinib combined with trastuzumab for maintenance therapy after first-line TH (P) therapy for HER2+ABC

DETAILED DESCRIPTION:
In this study, after at least 4 cycles of taxoid chemotherapy combined with trastuzumab ± pertuzumab, the evaluation result reached SD, CR or PR, and capecitabine combined with pyrotinib + trastuzumab was given successively in the later period (capecitabine was used for 4-6 cycles; Single-arm, multicenter, real-world observational studies using endocrine therapy + pyrrotinib + trastuzumab in patients with HR+, and maintenance therapy after first-line TH (P) therapy for CNS events (if non-CNS recurrent, progressive events occur and the investigator decides to change the follow-up regimen). To evaluate the effect of pyrrotinib combined with trastuzumab in maintaining treatment phase delay/reduction of brain metastases after first-line TH (P) therapy for advanced breast cancer with HER-2 positivity, the incidence of first progression of brain metastases was used as the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-70 years old, female;
2. Pathological examination confirmed HER-2 positive invasive breast cancer; Her2-positive is defined as >10% of tumor cells with an immunohistochemical (IHC) score of 3+ or in situ hybridization (ISH) results as HER2 gene amplification. A positive HER2 should be confirmed by the pathology department of the participating center of this study.) Imaging examination confirmed recurrent/metastatic breast cancer;
3. Patients with recurrence or metastasis more than 1 year after trastuzumab treatment, or newly diagnosed stage IV breast cancer;
4. ECOG score is 0-1;
5. Expected survival ≥6 months;
6. Normal function of major organs;
7. 1) Blood routine • ANC≥1.5×109/L; • PLT≥90×109/L; • Hb≥90 g/L; 2) Blood biochemistry • TBIL≤1.5×ULN; • ALT and AST≤2 x ULN; For patients with liver metastases, ALT and AST≤5× ULN; • BUN and Cr ≤ 1.5×ULN and creatinine removal rate ≥ 50 mL/min; 3) Heart color ultrasound • LVEF≥50%;
8. The researcher believes that the subject is likely to benefit;
9. Voluntarily participate in the study and sign the informed consent

Exclusion Criteria:

1. Head MRI or head CT confirms the presence of brain metastases;
2. Have multiple factors affecting oral medication (history of gastrointestinal surgery, inability to swallow, chronic diarrhea, intestinal obstruction);
3. Study patients allergic to drugs and excipients;
4. Suffering from mental illness or psychotropic substance abuse, unable to cooperate;
5. Pregnant or lactating women;
6. Participated in clinical trials within 4 weeks;
7. Participants considered unsuitable for inclusion by the researchers.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HER2-positive ABC
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of brain metastases | through study completion, an average of 2 year
  Incidence of brain metastases at first disease progression

SECONDARY OUTCOMES:
ORR | 24 month
  Overall Response Rate
PFS | through study completion, an average of 2 year
  Progression-free survival
OS | through study completion, an average of 3 year
  overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Union Medical College Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No